CLINICAL TRIAL: NCT07302321
Title: Investigation Into the Needs of ALS Patients With C9orf72 Mutation and Their Caregivers
Brief Title: Needs of ALS Patients With C9orf72 Mutation and Their Caregivers
Acronym: C9survALS
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 23C510
Record Dates: First submitted 2025-11-28; First posted 2025-12-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; C9orf72 mutation; Quality of life; Social Care Needs; Caregiver
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Surveys and Questionnaires; Caregivers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALS Patients with C9orf72 Mutation: Survey to describe the various aspects related to the care, needs and quality of life of C9orf72 ALS patients
  Interventions: Other: Survey for ALS patients
- Caregivers: Survey to describe the various aspects related to the care and time commitment for the assistance given by caregivers to C9orf72 ALS patients
  Interventions: Other: Survey for Caregivers

INTERVENTIONS:
Other: Survey for ALS patients — Survey to describe the various aspects related to the care, needs and quality of life of C9orf72 ALS patients
  Groups: ALS Patients with C9orf72 Mutation
Other: Survey for Caregivers — Survey to describe the various aspects related to the care and time commitment for the assistance given by caregivers to C9orf72 ALS patients
  Groups: Caregivers

SUMMARY:
Individuals with Amyotrophic Lateral Sclerosis (ALS) carrying the C9orf72 HRE mutation (C9Pos) often exhibit different phenotypic traits compared to other patients (C9Neg), presenting a more aggressive form of the disease, with also a higher frequency of comorbidity with frontotemporal dementia (ALS-FTD) and a greater prevalence of family history of ALS and/or other neurodegenerative diseases.

Considering these characteristics (comorbidity with FTD and family history of ALS and/or other neurodegenerative pathologies) as factors that have their importance from an assistance point of view, both C9orf72 patients and their caregivers may have particular needs in several respects, and in this sense this investigation is configured.

This survey aims to describe the various aspects related to the care and quality of life of C9orf72 ALS patients and their respective caregivers, with the goal of identifying actionable steps to improve the quality of life for both.

ELIGIBILITY:
ALS Patients:

Inclusion Criteria:

* Diagnosis of ALS with mutation C9orf72 (C9Pos)
* Age 18 years or older
* Fluency in Italian language
* Ability to understand the nature of the study and to reply to the questions in the online survey
* Informed consent signed

Exclusion Criteria:

* Clinically relevant cognitive dysfunction
* Incapacity to reply to at least half of the questions of the online survey
* Hospital Anxiety and Depression Scale (HADS) ≥ 11

Caregivers:

Inclusion Criteria:

* Caregiver of patient with diagnosis of ALS with mutation C9orf72 (C9Pos), who participates in this study
* Age 18 years or older
* Preserved cognitive functions
* Informed consent signed

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ALS patients with mutation C9orf72 (C9Pos) and their caregivers
Sampling Method: Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Multidisciplinary care | At enrolment
  ALS Patients with C9orf72 Mutation: Percentage with Multidisciplinary care
Home care | At enrolment
  ALS Patients with C9orf72 Mutation: Percentage with Home care
Satisfaction of primary needs | At enrolment
  ALS Patients with C9orf72 Mutation: Percentage with Satisfaction of primary needs
Satisfaction of economic support | At enrolment
  ALS Patients with C9orf72 Mutation: Percentage with Satisfaction of economic support
Age | At enrolment
  Caregivers: Age
Burdensome commitment | At enrolment
  Caregivers: Percentage of caregivers who perceive the assistance as a Burdensome commitment
Psychological support | At enrolment
  Caregivers: Percentage of caregivers who makes use of Psychological support

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Istituto Auxologico Italiano IRCCS, Milan, Lombardy
  - IRCCS Ospedale San Raffaele, Milan
  - IRCCS Fondazione Mondino, Istituto Neurologico Nazionale a Carattere Scientifico, Pavia